CLINICAL TRIAL: NCT05152797
Title: Efficacy and Safety of Autologous Tumor-infiltrating Lymphocytes in Treatment of Patients With Advanced or Metastatic Refractory Gynecological Cancer: a Prospective Multicenter One-arm Phase Ⅱ Trial
Brief Title: Efficacy and Safety of TILs in Treatment of Patients With Advanced or Metastatic Refractory Gynecological Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Tongji Hospital (Other); Qilu Hospital of Shandong University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO2021-1428
Record Dates: First submitted 2021-11-28; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Tumor Infiltrating Lymphocytes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TILs infusion (Experimental): Enrolled patients will be infused with their autologous TILs followed by IL-2 administration after post- NMA lymphodepletion
  Interventions: Biological: Autologous tumor-infiltrating lymphocytes

INTERVENTIONS:
Biological: Autologous tumor-infiltrating lymphocytes — Fresh tumor samples will be resected from enrolled patients. Autologous TILs will be extracted and reinfused to corresponding patients after ex vivo stimulation, activation and extensive expansion.

SUMMARY:
Prospective, multicenter, single-arm, open label, interventional basket trial to evaluate autologous tumor-infiltrating lymphocytes (TILs) infusion followed by IL-2 after a non-myeloablative (NMA) lymphodepletion preparation for the treatment of patients with advanced or metastatic refractory gynecological cancer including cervical, ovarian, endometrial and breast carcinoma.

DETAILED DESCRIPTION:
Autologous tumor-infiltrating lymphocytes (TILs) infusion is highly personalized cancer immunotherapy with strong anti-tumor efficacy and tumor specificity. TILs were extracted from autologous fresh tumor tissues, and after ex vivo stimulation, activation and extensive expansion, are reinfused to patients. TIL-based therapies have only been offered in small phase I/II studies in a few centers and revealed a high objective response rate (ORR) in the treatment of metastatic, recurrent or advanced melanoma, non-small cell long carcinoma and cervical carcinoma. However, the efficacy of TIL-based therapies still needs more clinical trials to prove. In this proposal, a one-arm, open, multicenter, phaseⅠ/Ⅱ trial was designed to evaluate the efficacy and safety of autologous tumor-infiltrating lymphocytes in treatment of patients with advanced or metastatic refractory gynecological cancer including cervical, ovarian, endometrial and breast carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this study must meet all of the following criteria: Signed informed consent must be obtained prior to participation in the study.

* Aged 18-75 years old at the time of consent
* Participants are diagnosed with advanced or metastatic cervical cancer, ovarian cancer, endometrial cancer or breast cancer with radiology and pathology confirmation.
* Failure of two or more Lines of Chemotherapy, or not amenable to curative treatment.
* At least one resectable lesion (or aggregate of lesions resected) of a minimum 1.5 cm in diameter post-resection to extract TIL
* At least one measurable target lesion, that can be accurately measured in at least one dimension with longest diameter ≥20 mm, as defined by RECIST v1.1
* All the chemotherapy or radiotherapy targeting the malignant tumors must be discontinued at least 28 days prior to the tumor resection.
* No serious abnormality of complete blood count and Cardiac, Liver, and Kidney function

Exclusion Criteria:

* Participants who have received organ transplantation or prior cell transfer therapy
* Any active autoimmune disease or history of autoimmune disease, or history of primary immunodeficiency.
* Patients who are taking systemic steroid therapy
* Patients with confirmed HIV infection, or other uncontrolled active viral infections, or serious system infections
* Patients with serious complications of heart, lung, liver, kidney, not suitable for enrollment.
* Patients with suspicious or confirmed brain metastases of any size and any number.
* Suffered from any other malignancy within 5 years (except for fully treated in situ malignant such as breast cancer, bladder cancer, cutaneous basal cell carcinoma or squamous cell carcinoma)
* Patients who are pregnant or breastfeeding
* Any other conditions judged by the researcher will significantly increase the risk of participation.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 6 months
  To evaluate the efficacy of TILs in patients with advanced or metastatic refractory malignant gynecological cancer including cervical, ovarian, endometrial and breast carcinoma based on the objective response rate (ORR) as assessed by the Independent Review Committee (IRC) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Disease Control Rate | Up to 60 months
  To evaluate the efficacy of TILs in patients with advanced or metastatic refractory gynecological cancer including cervical, ovarian, endometrial and breast carcinoma based on the disease control rate (DCR) as assessed by the IRC per RECIST v1.1
Progression-Free Survival | Up to 60 months
  To evaluate the efficacy of TILs in patients with advanced or metastatic refractory gynecological cancer including cervical, ovarian, endometrial and breast carcinoma based on the progression-free survival (PFS) as assessed by the IRC per RECIST v1.1
Overall Survival | Up to 60 months
  To evaluate overall survival (OS) in patients with advanced or metastatic refractory gynecological cancer including cervical, ovarian, endometrial and breast carcinoma
Adverse Events | Up to 60 months
  To characterize the safety profile of TILs in patients with advanced or metastatic refractory gynecological cancer including cervical, ovarian, endometrial and breast carcinoma as assessed by incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wang, MD, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University

IPD SHARING:
Plan to Share IPD: No